CLINICAL TRIAL: NCT02658994
Title: Thinking Healthy Program - Peer Delivered in Pakistan - Child-Focused
Brief Title: Thinking Healthy Program Peer Delivered Plus
Acronym: THPP+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Human Development Research Foundation, Pakistan (Other)
Collaborators: Duke University (Other); Columbia University (Other); University of Liverpool (Other); University of Essex (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: THPPPlusChild001
Record Dates: First submitted 2016-01-13; First posted 2016-01-20 (Estimated); Results first posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- THPP+ (Experimental): As part of THPP+, the intervention will continue from the 6th month postnatal through 36 months postnatal and so will consist of an additional 30 months of lower intensity services that are unique to THPP+. The THPP+ will also include additional group sessions to be held every other month for a total of 18 over the intervention duration. The content will be a continuation of the previous THPP sessions with continuing emphasis on self-care as well as the baby's health and development.
  Interventions: Behavioral: Thinking Healthy Program Peer Delivered Plus
- Enhanced Usual Care (Active Comparator): Women in the control clusters who were depressed prenatally have been receiving Enhanced Usual Care (EUC). At the time of the screening, women, their Lady Health Workers, and their local primary health care facility were informed of the diagnosis, and women were given an information sheet about depression and how to access care. There are no new EUC protocols put in place post-partum as part of the THPP+.
  Interventions: Other: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Thinking Healthy Program Peer Delivered Plus
  Arms: THPP+
Other: Enhanced Usual Care
  Arms: Enhanced Usual Care

SUMMARY:
Background

The negative effects of perinatal depression on mother and child start early and persist throughout the life-course. Given that 10-35% of children worldwide are exposed to perinatal depression in their first year of life, 16 mitigating this intergenerational risk is a global public health priority. However, there is a dearth of studies on whether a maternal depression intervention can have long-term benefits for either the mother or her child. This is a study of the effectiveness of an extended 36-month peer-delivered depression intervention, the Thinking Healthy Programme PLUS (THPP+) for women and their children in rural Pakistan.

Study Design

The THPP+ study aims to evaluate the effects of an extended 36-month perinatal depression intervention on mother and child outcomes using a cluster randomized controlled trial (c-RCT) design. The trial will recruit 560 pregnant women who screened positive for perinatal depression (PHQ-9 >=10) from 40 village clusters, of which 20 clusters will receive the THPP+ intervention delivered by trained peers. These women will have already been participating in the trial of the shorter, 6 month long, version of the intervention. Women in the THPP+ intervention arm will receive bimonthly group-based sessions. Primary outcomes are 3-year maternal depression and 3-year child socio-emotional and cognitive development. All primary analyses will be intention-to-treat and will account for the clustered study design.

Discussion

This trial has the potential to further significantly our understanding of whether intervening on women's perinatal depression can mitigate the negative effects of maternal depression on 36-month child development.

DETAILED DESCRIPTION:
Every year millions of children begin a compromised developmental trajectory resulting from exposure to maternal depression. In recent years, compelling evidence that maternal depression leads to worse developmental outcomes in the child has prompted a dramatic increase in efforts to ameliorate it. However, empirical evidence linking depression treatment to improved developmental trajectories in offspring is far from robust. The evidence is lacking due to several methodological limitations of previous studies, namely, insufficient follow-up, lack of appropriate control group, and/or lack of attention to the psychological and behavioral mechanisms underlying the impact of interventions on both the mother and child.

We propose an innovative, cost-effective extension to an NIMH-funded perinatal depression cluster randomized controlled intervention trial (RCT) in Pakistan (SHARE: U19MH095687). The SHARE RCT includes individual and community-wide components and follows mothers with prenatal depression until 6 months postpartum. Our proposal, SHARE CHILD, builds on this trial in several critical ways. We (1) focus on child outcomes, (2) extend follow-up to 36 months postpartum, (3) include mothers who did not screen positive for depression in the 3rd trimester, thus enabling additional comparisons, and (4) investigate factors that mediate and modify the effect of the intervention on child outcomes. A unique window of opportunity is made possible due to the anticipated spring 2014 enrollment start date of the SHARE trial.

Our long-term goal is to identify key modifiable factors in the intergenerational transmission of risk from depressed mothers to their children. The overall objective of this proposal is to rigorously evaluate the impact of a community based perinatal depression intervention on child development by expanding the sample of an already funded RCT and extending the follow-up period to 36 months postpartum. Our central hypothesis is that the perinatal depression intervention will lead to improved child socio-emotional, cognitive, and physical outcomes. Including the non-depressed dyads in our analyses will enable us to further determine (a) how much of the excess risk due to maternal depression exposure the intervention can mitigate and (b) whether this community based intervention has an impact on all children living in the intervention clusters, even if their mothers were not depressed prenatally. Such insights would not otherwise be possible without this expanded sample given the dearth of information on child developmental norms in this setting. Together, the unique opportunity to extend the SHARE trial to the broader SHARE CHILD study and the approaches we propose will yield novel and definitive evidence of the impact of treating perinatal depression on child developmental outcomes.

ELIGIBILITY:
Inclusion Criteria:

* currently enrolled in THPP trial
* married
* residing in study area for the long term

Exclusion Criteria:

* Requiring immediate medical attention
* development of psychotic or manic episode
* broken mother-child dyad

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1154 (Actual)
Dates: Start 2014-10; Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Siham Sikander, Principal Investigator — Human Development Research Foundation, Pakistan
Locations (1):
- Human Development Research Foundation, Islamabad, Pakistan

REFERENCES:
- [Derived] LeMasters K, Bates LM, Chung EO, Gallis JA, Hagaman A, Scherer E, Sikander S, Staley BS, Zalla LC, Zivich PN, Maselko J. Adverse childhood experiences and depression among women in rural Pakistan. BMC Public Health. 2021 Feb 25;21(1):400. doi: 10.1186/s12889-021-10409-4. PMID 33632175
- [Derived] Maselko J, Sikander S, Turner EL, Bates LM, Ahmad I, Atif N, Baranov V, Bhalotra S, Bibi A, Bibi T, Bilal S, Biroli P, Chung E, Gallis JA, Hagaman A, Jamil A, LeMasters K, O'Donnell K, Scherer E, Sharif M, Waqas A, Zaidi A, Zulfiqar S, Rahman A. Effectiveness of a peer-delivered, psychosocial intervention on maternal depression and child development at 3 years postnatal: a cluster randomised trial in Pakistan. Lancet Psychiatry. 2020 Sep;7(9):775-787. doi: 10.1016/S2215-0366(20)30258-3. PMID 32828167
- [Derived] LeMasters K, Andrabi N, Zalla L, Hagaman A, Chung EO, Gallis JA, Turner EL, Bhalotra S, Sikander S, Maselko J. Maternal depression in rural Pakistan: the protective associations with cultural postpartum practices. BMC Public Health. 2020 Jan 15;20(1):68. doi: 10.1186/s12889-020-8176-0. PMID 31941468
- [Derived] Scherer E, Hagaman A, Chung E, Rahman A, O'Donnell K, Maselko J. The relationship between responsive caregiving and child outcomes: evidence from direct observations of mother-child dyads in Pakistan. BMC Public Health. 2019 Feb 28;19(1):252. doi: 10.1186/s12889-019-6571-1. PMID 30819173
- [Derived] Turner EL, Sikander S, Bangash O, Zaidi A, Bates L, Gallis J, Ganga N, O'Donnell K, Rahman A, Maselko J. The effectiveness of the peer delivered Thinking Healthy Plus (THPP+) Programme for maternal depression and child socio-emotional development in Pakistan: study protocol for a three-year cluster randomized controlled trial. Trials. 2016 Sep 8;17(1):442. doi: 10.1186/s13063-016-1530-y. PMID 27608926

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1154 pregnant women were enrolled in the study. Enhanced usual care (EUC) group had 287, THPP had 283, no prenatal depression had 584. The study team attempted to interview all women at all follow up visits (baseline, 3 mo, 6 mo, 12 mo, 24 mo, 36 mo). If a woman missed a previous visit, (LTFU, temporarily absent, refused) she was not excluded from participating in further visits. Therefore, the number of participants at each follow up visit may increase and decrease but will not exceed 1154.
Groups:
- THPP+: As part of THPP+, the intervention will continue from the 6th month postnatal through 36 months postnatal and so will consist of an additional 30 months of lower intensity services that are unique to THPP+. The THPP+ will also include additional group sessions to be held every other month for a total of 18 over the intervention duration. The content will be a continuation of the previous THPP sessions with continuing emphasis on self-care as well as the baby's health and development.
  Thinking Healthy Program Peer Delivered Plus
- No Prenatal Depression: No prenatal depression recorded at baseline.
Period: Enrollment
Arm/Group | Enhanced Usual Care | THPP+ | No Prenatal Depression
Started | 287 | 283 | 584
Completed | 287 | 283 | 584
Not Completed | 0 | 0 | 0
Period: 3 Month Follow up
Arm/Group | Enhanced Usual Care | THPP+ | No Prenatal Depression
Started | 287 | 283 | 584
Completed | 221 | 223 | 451
Not Completed | 66 | 60 | 133
Period: 6 Month Follow up
Arm/Group | Enhanced Usual Care | THPP+ | No Prenatal Depression
Started | 287 (Participants who did not complete 3 month follow up were still eligible for 6 month follow up) | 283 (Participants who did not complete 3 month follow up were still eligible for 6 month follow up) | 584 (Participants who did not complete 3 month follow up were still eligible for 6 month follow up)
Completed | 228 | 230 | 471
Not Completed | 59 | 53 | 113
Period: 12 Month Follow up
Arm/Group | Enhanced Usual Care | THPP+ | No Prenatal Depression
Started | 287 (Participants who did not complete 6 month follow up were still eligible for 12 month follow up) | 283 (Participants who did not complete 6 month follow up were still eligible for 12 month follow up) | 584 (Participants who did not complete 6 month follow up were still eligible for 12 month follow up)
Completed | 228 | 223 | 489
Not Completed | 59 | 60 | 95
Period: 24 Month Follow up
Arm/Group | Enhanced Usual Care | THPP+ | No Prenatal Depression
Started | 287 (Participants who did not complete 12 month follow up were still eligible for 24 month follow up) | 283 (Participants who did not complete 12 month follow up were still eligible for 24 month follow up) | 584 (Participants who did not complete 12 month follow up were still eligible for 24 month follow up)
Completed | 220 | 210 | 473
Not Completed | 67 | 73 | 111
Period: 36 Month Follow up
Arm/Group | Enhanced Usual Care | THPP+ | No Prenatal Depression
Started | 287 (Participants who did not complete 24 month follow up were still eligible for 36 month follow up) | 283 (Participants who did not complete 24 month follow up were still eligible for 36 month follow up) | 584 (Participants who did not complete 24 month follow up were still eligible for 36 month follow up)
Completed | 216 | 206 | 467
Not Completed | 71 | 77 | 117

BASELINE CHARACTERISTICS:
Groups:
- Enhanced Usual Care: Informing participants and LHWs about depression status and ways to seek help.
- THPP and THPP+: Group based booster sessions which included peer support behavioral activation and problem solving.
- No Prenatal Depression: No prenatal depression at baseline.
- Total: Total of all reporting groups
Arm/Group | Enhanced Usual Care | THPP and THPP+ | No Prenatal Depression | Total
Number analyzed (Participants) | 287 | 283 | 584 | 1154
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 287 | 283 | 584 | 1154
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 287 | 283 | 584 | 1154
  Male | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Pakistan | 287 | 283 | 584 | 1154
Mother's education [Count of Participants; unit: Participants]
  None | 55 | 52 | 63 | 170
  Primary (1-5) | 71 | 68 | 87 | 226
  Middle or secondary (6-12) | 134 | 145 | 338 | 617
  Tertiary >13 | 27 | 18 | 96 | 141
Nuclear family [Count of Participants; unit: Participants] — Nuclear family describes the household composition. Nuclear family is a two parent household.
  Participants | 49 | 50 | 59 | 158
Total number of children in the household [Count of Participants; unit: Participants]
  First pregnancy | 72 | 65 | 212 | 349
  1-3 | 183 | 180 | 336 | 699
  4 or more | 32 | 38 | 36 | 106
Duration of depression (chronicity) [Count of Participants; unit: Participants] — Population: This group did not have prenatal depression at baseline.
  Participants
    number analyzed (Participants) | 287 | 283 | 0 | 570
    <12 weeks | 38 | 35 |  | 73
    >12 weeks | 155 | 171 |  | 326
    Data missing | 94 | 77 |  | 171
SES (assets) [Count of Participants; unit: Participants]
  Lowest quintile | 74 | 85 | 71 | 230
  Lower-middle quintile | 67 | 71 | 93 | 231
  Middle quintile | 55 | 50 | 126 | 231
  Upper-middle quintile | 47 | 39 | 145 | 231
  Upper quintile | 44 | 38 | 149 | 231

OUTCOME MEASURES:

1. Primary Outcome: Depression (PHQ-9 Instrument)
Description: The PHQ-9 is a 9-question instrument given to patients in a primary care setting to screen for the presence and severity of depression. The results may be used to make a depression diagnosis according to the DSM-IV criteria. The PHQ-9 asks about patients experience in the last two weeks. Questions are about the level of interest in doing things, feeling down or depressed, difficulty with sleeping, energy levels, eating habits, self-perception, ability to concentrate, speed of functioning and thoughts of suicide. Responses range from "0" (not at all) to "3" (nearly every day). Scores range from 0-27, a total of 10 or above is suggestive of the presence of depression.
  PHQ-9 score Depression severity 0-4 minimal depression 5-9 mild depression 10-14 moderate depression 15-19 moderately severe depression 20+ severe depression
Time Frame: 36 months post-partum
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced Usual Care | THPP and THPP+ | No Prenatal Depression
Number analyzed (Participants) | 216 | 206 | 467
score on a scale | 6.48 (6.25) | 5.84 (5.80) | 3.44 (4.53)
Statistical Analysis 1: Comparison: Enhanced Usual Care vs THPP and THPP+; Test type: Superiority; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-0.33 to 0.07]

2. Primary Outcome: Child Strength and Difficulties Questionnaire (SDQ) Total Difficulties (TD) Score
Description: The SDQ is a parent-reported measure of 25 child attributes with five subscales of 5 items each; emotional symptoms, conduct problems, hyperactivity, peer problems, and prosocial behavior. The TD score is calculated on the basis of four subscales (omitting prosocial behavior) with a score range of 0-40 points. The SDQ is widely used in low and middle-income countries and has been translated into Urdu. High SDQ scores are associated with a substantial increase in psychiatric risk.
  The TD score of our child participants is listed as a mean in the values below. TD score of 0-13 is considered "close to average, clinically significant problems in this area are unlikely," 14-16 is "slightly raised, which may reflect clinically significant problems," and 17-40 is "high, there is substantial risk of clinically significant problems in this area."
Time Frame: 36 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced Usual Care | THPP and THPP+ | No Prenatal Depression
Number analyzed (Participants) | 216 | 206 | 467
score on a scale | 14.72 (6.13) | 14.73 (6.04) | 13.69 (6.34)
Statistical Analysis 1: Comparison: Enhanced Usual Care vs THPP and THPP+; Test type: Superiority; Median Difference (Final Values) = -0.10, 95% CI 2-sided [-1.39 to 1.19]

3. Secondary Outcome: Disability (WHO Disability Assessment Schedule 2.0)
Description: WHODAS 2.0 was used to assess disability in the women in the cohort, the 12-item questionnaire was used to assess level of functionality over the last 30 days. The cohort was asked questions 2-13, and simple scoring was used. Responses to questions were none (0 points), mild difficulty (1 point), severe difficulty (2 points), and extreme difficulty/cannot do (4 points). Responses to the items were summed and scaled to a 0-100 scale to compute a total score, where 0 indicated no disability and 100 indicated full disability.
Time Frame: 36 months post-partum
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced Usual Care | THPP and THPP+ | No Prenatal Depression
Number analyzed (Participants) | 216 | 206 | 467
score on a scale | 16.11 (9.12) | 16.71 (8.52) | 5.61 (6.46)
Statistical Analysis 1: Comparison: Enhanced Usual Care vs THPP and THPP+; Test type: Superiority; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-0.33 to 0.09]

4. Secondary Outcome: Infant Cognitive Development (Bayley Scales of Infant Development)
Description: Bayley Scales of Infant Development-III (BSITD) is an individually administered assessment of the child's achievement of developmental milestones across five areas. For this study, we focus on receptive language and fine motor domains at 36 months. A higher score means higher functioning. The two subscales are not combined, but treated as separate variables. The subscales are scaled according to the procedure outlined in the Bayley reference manual, the scaled score minimum and maximums at 36 months are: Receptive- min: 5; max: 19, Fine Motor- min: 2; max: 19.
Time Frame: 36 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced Usual Care | THPP and THPP+ | No Prenatal Depression
Number analyzed (Participants) | 216 | 206 | 467
score on a scale
  Child Bayley scaled receptive score | 9.98 (2.60) | 10.42 (2.81) | 10.41 (2.79)
  Child Bayley scaled fine motor score | 11.38 (4.12) | 11.42 (4.05) | 11.31 (3.99)
Statistical Analysis 1: Comparison: Enhanced Usual Care vs THPP and THPP+; Child Bayley scaled receptive score; Test type: Superiority; Mean Difference (Final Values) = 0.38, 95% CI 2-sided [-0.19 to 0.96]
Statistical Analysis 2: Comparison: Enhanced Usual Care vs THPP and THPP+; Child Bayley scaled fine motor score; Test type: Superiority; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.83 to 0.90]

5. Secondary Outcome: Number of Participants With Depression (SCID Major Depressive Episode)
Description: SCID is a semi-structured interview for the diagnoses of psychiatric disorders. It has been cross-culturally adapted for assessing depression among women during pregnancy and in the postpartum period. The PHQ-9 inquires about frequency of depressive symptoms in the last 2 weeks. Given that the PHQ-9 is a screening tool, we use the SCID module for current major depressive episode as a diagnostic tool to assess the criterion-related validity of using the scores from the PHQ-9 to measure the number of symptoms endorsed by the woman over time. The diagnostic and statistical manual of mental disorders (DSM) IV diagnosis of current major depressive episode is generated through the SCID algorithm. If a woman was diagnosed with at least 1 MDE she was included in the outcome below.
Time Frame: 36 months post-partum
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Usual Care | THPP and THPP+ | No Prenatal Depression
Number analyzed (Participants) | 216 | 206 | 467
Participants | 48 | 34 | 42
Statistical Analysis 1: Comparison: Enhanced Usual Care vs THPP and THPP+; Test type: Superiority; Risk Ratio (RR) = 0.67, 95% CI 2-sided [0.43 to 1.05]

6. Other Pre Specified Outcome: Infant Physical Development [Z-scores (Based on WHO Criteria)]
Description: Child growth was analyzed with the weight-for-age and length-for-age z scores.
Time Frame: 36 months
Measure: Mean (Standard Deviation); unit: z score
Arm/Group | Enhanced Usual Care | THPP and THPP+ | No Prenatal Depression
Number analyzed (Participants) | 216 | 206 | 467
z score
  length-for-age | -1.03 (1.01) | -1.12 (1.13) | -0.96 (1.11)
  weight-for-age | -0.95 (1.03) | -1.06 (0.97) | -0.94 (0.98)
Statistical Analysis 1: Comparison: Enhanced Usual Care vs THPP and THPP+; Length-for-age z-scores; Test type: Superiority; Risk Ratio (RR) = -0.09, 95% CI 2-sided [-0.32 to 0.15]
Statistical Analysis 2: Comparison: Enhanced Usual Care vs THPP and THPP+; Weight-for-age z-scores; Test type: Superiority; Risk Ratio (RR) = -0.12, 95% CI 2-sided [-0.33 to 0.10]

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 3 years
Arm/Group | Enhanced Usual Care | THPP and THPP+ | No Prenatal Depression
All-Cause Mortality (participants affected / at risk) | 30/287 | 28/283 | 47/584
Serious Adverse Events (participants affected / at risk) | 0/287 | 0/283 | 0/584
Other Adverse Events (participants affected / at risk) | 3/287 | 5/283 | 7/584
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enhanced Usual Care (N=287) | THPP and THPP+ (N=283) | No Prenatal Depression (N=584)
Hernia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Child illness (General disorders) | 3 (3) | 4 (4) | 4 (4)
Mother illness (General disorders) | 0 (0) | 1 (1) | 1 (1)
Child disability (General disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The indicators of child socioemotional outcomes, although measured with validated and extensively used instruments, were mother reported, and, as such, susceptible to bias. However, if depression symptoms biased reporting, we would expect this to have affected the overall socioemotional domain, not just the hyperactivity or conduct problems reported in our study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-04-15): https://cdn.clinicaltrials.gov/large-docs/94/NCT02658994/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-14): https://cdn.clinicaltrials.gov/large-docs/94/NCT02658994/SAP_001.pdf